CLINICAL TRIAL: NCT03591367
Title: The Potential Role Of MicroRNA-155 And Telomerase Reverse Transcriptase In Diagnosis Of Non-Muscle Invasive Bladder Cancer And Their Pathological Correlation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MicroRNA-155 Bladder Cancer
Record Dates: First submitted 2018-07-08; First posted 2018-07-19 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2018-07

CONDITIONS: Bladder Cancer; Bladder Disease; Bladder Neoplasm; Micro-RNA
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urinary Bladder Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hematuria due to suspicious superficial bladder tumor (Other): MicroRNAs-155 (miRNAs-155) and Human telomerase reverse transcriptase (hTERT)
  Interventions: Diagnostic Test: MicroRNAs-155; Diagnostic Test: Human telomerase reverse transcriptase

INTERVENTIONS:
Diagnostic Test: MicroRNAs-155 — Quantitative analysis of cell-free miR-155 using RT-qPCR.
  Other Names: (miRNAs-155)
Diagnostic Test: Human telomerase reverse transcriptase — Analysis TERT by TERT messenger RNA (mRNA)expression by reverse transcription-quantitative polymerase chain reaction.
  Other Names: (hTERT)

SUMMARY:
We try to assess the potential role of telomerase reverse transcriptase and MicroRNA (miR-155) in diagnosis of non-muscle-invasive bladder cancer and their correlation with stage and grade of the tumor.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years or older.
* Patient with hematuria suspected to be of bladder origin clinically.
* Willing to be participate in the study.

Exclusion Criteria:

* Patient having another malignancy.
* Hematuria of other causes as trauma and stones

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
sensitivity, specificity and positive and negative predictive values of combined MicroRNA-155 And Telomerase Reverse Transcriptase In diagnosis Of Non-Muscle Invasive Bladder Cancer | 1 year
  compared by standard final pathological specimen

SECONDARY OUTCOMES:
correlation between serum Vit D and Non-Muscle Invasive Bladder Cancer | 1 year
  measured serum Vit D in ng/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mosbah, MD, Study Chair — Urology and nephrology center
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Aldakahlia, Egypt